CLINICAL TRIAL: NCT04906928
Title: Evaluation of the Performance of a 3D FGAPSIR Sequence by MRI in the Detection and Characterization of Spinal Cord Injuries in Patients With Multiple Sclerosis
Brief Title: Evaluation of New MRI Sequences Including 3D-FGAPSIR for the Optimization of Inflammatory Spinal Cord Lesions Research
Acronym: ESPOIR2
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2021_15
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — * standard imaging protocol prescribed as part of the usual treatment: sagittal T1 and T2 slices after injection of contrast product (Gadolinium), 3D STIR and 3D PSIR sequence.
  * 3D FGAPSIR sequence at the level of the cervical cord for the duration of the additional sequence is 10 minutes, for a total examination time of 40 minutes (instead of 30 minutes)

SUMMARY:
* verification of inclusion and non-inclusion criteria
* information and collection of consent
* standard imaging protocol prescribed as part of the usual treatment: sagittal T1 and T2 slices after injection of contrast product (Gadolinium), 3D STIR and 3D PSIR sequence.
* 3D FGAPSIR sequence at the level of the cervical cord for the duration of the additional sequence is 10 minutes, for a total examination time of 40 minutes (instead of 30 minutes)

DETAILED DESCRIPTION:
* verification of inclusion and non-inclusion criteria
* information and collection of consent
* standard imaging protocol prescribed as part of the usual treatment: sagittal T1 and T2 slices after injection of contrast product (Gadolinium), 3D STIR and 3D PSIR sequence.
* 3D FGAPSIR sequence at the level of the cervical cord for the duration of the additional sequence is 10 minutes, for a total examination time of 40 minutes (instead of 30 minutes)

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* To benefit from a medullary exploration planned by 3T MRI as part of a first evaluation or a reassessment of inflammatory involvement of the nevrax
* Express consent to participate in the study
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant, parturient or breastfeeding woman
* Absolute or relative contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be offered prospectively to patients presenting to the imaging department for a 3T MRI for bone marrow exploration, in the context of inflammatory involvement of the nevrax
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
estimate the number of lesions detected with the 3D FGAPSIR sequence and not detected with the 3D PSIR sequence. | 1 DAY
  estimate the number of lesions detected with the 3D FGAPSIR sequence and not detected with the 3D PSIR sequence.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild (FOR), Paris, France